CLINICAL TRIAL: NCT07065695
Title: A Prospective Randomized Controlled Study on the Safety and Effectiveness of Microscopic Varicocele Bypass Surgery Compared With Simple Ligation
Brief Title: Microscopic Varicocele Bypass Versus Ligation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ke Dou (Other)
Responsible Party: Sponsor-Investigator, Ke Dou, Sichuan Provincial People's Hospital, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025358
Record Dates: First submitted 2025-05-30; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Varicocele
Keywords: Varicocele; microscopic simple ligation; transposition surgery
MeSH Terms: conditions — Varicocele

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transposition surgery (Experimental): Reconstructs spermatic vein drainage via end to end anastomosis with inferior epigastric vein
  Interventions: Procedure: transposition surgery
- simple ligation (Active Comparator): Blocks venous reflux via double ligation and division of spermatic veins under microscopy
  Interventions: Procedure: microscopic simple ligation

INTERVENTIONS:
Procedure: transposition surgery — Reconstructs spermatic vein drainage via end to side/end to end anastomosis with vessels (e.g., inferior epigastric vein) under 8-15× magnification, preserving testicular arteries/lymphatics.
  Arms: transposition surgery
Procedure: microscopic simple ligation — Blocks venous reflux via double ligation and division of spermatic veins under microscopy, with identical surgical exposure and vascular protection.
  Arms: simple ligation

SUMMARY:
This study, titled "A Prospective Randomized Controlled Study on the Safety and Efficacy of Microscopic Varicocele Transposition Surgery Compared with Simple Ligation," is conducted by the Urology and Andrology Department of Sichuan Provincial People's Hospital, with Dou Ke serving as the principal investigator. The research period spans from May 2025 to December 2027. It aims to compare the outcomes of microscopic varicocele transposition surgery and simple ligation in treating left varicocele through a prospective randomized controlled trial, focusing on postoperative recovery, complications, semen quality, and other aspects to provide evidence for clinical surgical selection.

A total of 284 male patients will be enrolled, meeting criteria including clinical diagnosis of varicocele with surgical indications, aged 18-60 years, willing to participate and signing informed consent, abnormal semen analysis related to varicocele, no severe organ dysfunction, and no relevant treatments affecting the condition in the past three months. Exclusions include secondary varicocele, severe genitourinary or systemic diseases, coagulation disorders, drug allergies, mental/cognitive impairments, and participation in other related clinical trials. The experimental group will receive microscopic varicocele transposition surgery, while the control group will undergo microscopic simple ligation. Primary evaluation indicators include changes in spermatic vein diameter, reflux velocity, and duration assessed by color Doppler ultrasound at 1, 3, and 6 months post-surgery (with additional measurements of anastomotic vessel diameter and flow velocity in the experimental group), as well as pre- and post-surgery (3 and 6 months) semen routine parameters. Secondary indicators surgical success rate, postoperative complication rate, changes in reproductive hormone levels, pain relief evaluated by VAS scale, and quality of life improvements via specific assessment tools. Complying with the Declaration of Helsinki and approved by the ethics committee, informed consent will be obtained from all participants. Study results will be disseminated through academic papers, conference presentations, clinical research reports, and patient-focused summaries to advance new treatment directions for varicocele and optimize clinical protocols.

DETAILED DESCRIPTION:
This prospective, single-blind, randomized controlled trial is conducted at the Urology and Andrology Center of Sichuan Provincial People's Hospital, led by Principal Investigator Dou Ke, to evaluate the safety and efficacy of microscopic varicocele transposition surgery compared with microscopic simple ligation for treating left varicocele. The study spans from May 2025 to December 2027.

1. Study Design Details

   Randomization Process:

   Utilizing a computer-generated random number table with a 1:1 allocation ratio, patients are assigned to either group. To ensure randomness, the randomization sequence is generated by an independent statistician not involved in patient enrollment or intervention delivery. Block randomization with block sizes of 4-8 will be employed to balance group sizes over time.

   Blinding Implementation:

   In this single-blind design, patients remain unaware of their group assignment throughout the study. To maintain blinding, patient identification codes are used instead of names during follow-up, and outcome assessors are trained to conduct evaluations without accessing group allocation information. Surgeons and researchers directly involved in the surgical procedures are aware of the group assignment for proper procedure execution.

   Surgical Techniques:

   Experimental Group: Under 8-15× microscopic magnification, the surgical team will perform end-to-side or end-to-end anastomosis of the spermatic vein with other vessels, typically the inferior epigastric vein. The surgical procedure includes meticulous dissection to isolate the spermatic vein while carefully preserving the testicular artery, lymphatic vessels, and nerve fibers. Specialized microsurgical instruments, such as microscissors with a tip diameter of 0.1-0.3 mm and 10-11-0 nylon sutures, are used for precise anastomosis.

   Control Group: Microscopic simple ligation involves double ligation and division of the spermatic veins. The surgical field exposure, including the incision size (usually 3-4 cm), and the method of protecting testicular vasculature and other structures, are kept identical to the experimental group to minimize confounding factors.
2. Measurement and Assessment Details

   Ultrasound Evaluation:

   Color Doppler ultrasound will be performed using high-resolution machines (e.g., with a probe frequency of 7-12 MHz) by experienced sonographers blinded to group assignment. For the experimental group, when assessing anastomotic vessel patency, the angle of insonation will be maintained at ≤60° to accurately measure blood flow velocity. Standardized scanning protocols will be followed, including specific patient positions (supine and standing) to detect varicocele reflux.

   Semen Analysis:

   Semen samples will be collected via masturbation after 2-7 days of sexual abstinence and analyzed within 1 hour at a certified andrology laboratory. Automated semen analyzers will be used to measure sperm concentration, motility, and morphology, while liquefaction time will be assessed visually. Quality control procedures, including periodic calibration of the analyzer and internal proficiency testing, are in place to ensure data reliability.
3. Statistical Considerations

   Sample Size Calculation:

   Based on a previous study reporting a 15% difference in primary outcome improvement between similar surgical methods, with 80% power and a two-sided significance level of 0.05, a total sample size of 284 patients (142 per group) was determined. Adjustments for potential dropout rates (estimated at 10%) have been incorporated.

   Missing Data Handling:

   For continuous variables with missing data, multiple imputation methods will be used, considering baseline characteristics and other relevant variables. For categorical data, the last observation carried forward approach may be applied depending on the nature of missingness.
4. Ethical and Safety Oversight

   Ethical Review:

   The study protocol has been reviewed and approved by the institutional ethics committee of Sichuan Provincial People's Hospital. An annual ethics review will be conducted to monitor any protocol deviations or emerging ethical issues.

   Safety Monitoring:

   An independent Data and Safety Monitoring Board (DSMB) will review interim safety data every 6 months. In case of a serious adverse event (SAE), such as testicular artery injury leading to ischemia, the DSMB can recommend immediate changes to the protocol, including halting the trial if necessary.
5. Dissemination Plan

In addition to publishing in peer-reviewed urology and andrology journals and presenting at national/international conferences, the study team will collaborate with patient advocacy groups to develop infographics and short videos summarizing the key findings. These materials will be made available on the hospital's official website and social media platforms to enhance patient education and awareness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with varicocele and meet the surgical indications
* Male patients aged between 18 and 60 years old
* Patients have the willingness to receive treatment, voluntarily participate in this study and sign the informed consent form
* Semen analysis reveals abnormalities associated with varicocele
* The patient has no severe dysfunction of vital organs and can tolerate surgery
* The patient has received no relevant treatment affecting varicocele or semen quality in the past three months

Exclusion Criteria:

* Secondary varicocele
* Complicated with other severe reproductive system diseases
* Suffering from severe systemic diseases, which may affect the surgical effect or prognosis
* Presence of coagulation dysfunction or taking medications that affect coagulation function
* Having a history of allergy to the drugs used in the surgery
* Having mental illness or cognitive impairment and being unable to cooperate to complete this study
* Having already participated in other relevant clinical trials.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since this study is aimed at patients with varicocele, only males will be included in the study.
Enrollment: 284 (Estimated)
Dates: Start 2025-07-22 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of the surgery | 1, 3, and 6 months postsurgery
  measuring vein diameter，anastomotic vessel patency and reflux duration by color Doppler ultrasound
Semen analysis | 1, 3, and 6 months postsurgery
  Semen Quality by semen analysis

SECONDARY OUTCOMES:
The incidence rate of postoperative complications | postsurgery (3, 6 months)
  Mainly include bleeding, testicular artery injury, scrotal hematoma and infection
Testicular volume | postsurgery (3, 6 months)
  Measure the size of the testicles by ultrasound
Testicular function | postsurgery (3, 6 months)
  Determination of serum sex hormones

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT07065695/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT07065695/ICF_001.pdf